CLINICAL TRIAL: NCT06296849
Title: Randomized Controlled Trial of Dyadic Financial Incentive Treatments for Dual Smoker Couples: Evaluation of Efficacy, Mechanisms, and Cost Effectiveness (1R01CA276594-01A1)
Brief Title: Dyadic Financial Incentive Treatments for Dual Smoker Couples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: McMaster University (Other); University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROJECT00007344
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Smoking, Cigarette
Keywords: smoking cessation; dual-smoker couples; behavioral economics; financial incentives
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No-FIT Treatment-as-Usual (TAU) Condition (No Intervention): Participants in the no-FIT control condition will not receive incentives.
- Single-Target FIT (SFIT) (Experimental): One couple member offered incentives. Targets in the SFIT condition will be offered financial incentives for biochemically verified abstinence ($200 at each of three follow-ups [1, 3, and 6 Month]).
  Interventions: Behavioral: Financial Incentive Treatment (FIT)
- Dyadic-FIT condition (DFIT) (Experimental): Both couple members offered incentives and tracked across 12 months. Both targets and partners will be offered financial incentives for abstinence. Thus, in this condition, the total financial incentives offered to the dyad are twice the amount as offered to participants in the SFIT condition.
  Interventions: Behavioral: Financial Incentive Treatment (FIT)

INTERVENTIONS:
Behavioral: Financial Incentive Treatment (FIT) — In the present study, the investigators will provide financial incentives of $200 for biochemically verified abstinence at each of three time points (1 month, 3 month, and 6 month) following baseline. Additionally, the investigators will provide a bonus of $200 for participants who demonstrate abstinence at each of the time points. This incentive value is consistent with recent research using macro-level financial incentives and incorporates both short-term and long-term incentives to shape behavior.
  Arms: Dyadic-FIT condition (DFIT); Single-Target FIT (SFIT)

SUMMARY:
Smokers partnered with other smokers (i.e., dual-smoker couples) represent ~2/3 of all smokers. Dual-smoker couples (DSCs) are less likely to try to quit smoking and more likely to relapse during a quit attempt, reducing overall smoking cessation rates and representing a high-risk clinical population. Despite their high prevalence and risk for persistent smoking, however, there are limited data on smoking cessation interventions among DSCs. Building on previous research that suggests a) financial incentive treatments (FITs) are effective at increasing quit rates and b) dyadic adaptations of FITs are feasible for implementation in DSCs, the proposed study will systematically two versions of FITs to enhance smoking cessation among DSCs. In addition to determining the efficacy of these dyadic FITs for smoking abstinence in DSCs, the investigators will consider the cost and cost effectiveness of each adaptation as well as mechanisms of change to inform future implementation research. The investigators will additionally consider secondary outcomes including abstinence during treatment and long-term abstinence maintenance after end of treatment.

The investigators will address these questions in a three-group randomized controlled trial (RCT). In all conditions, individuals who have smoking partners (i.e., targets) will receive usual care (combination fast and slow acting Nicotine Replacement Therapy + quitting resources). In two conditions, participants will receive incentives for abstinence at three time points (1, 3, and 6 months post-baseline). In the SFIT condition, only the target in a couple will be offered incentives; in the DFIT condition, both target and partner will be offered incentives. Primary efficacy outcome is % point-prevalence abstinence at 6 months post-baseline among targets. Secondary outcomes are point-prevalence abstinence at 1 and 3 months during the treatment and 6 months post-treatment (12-months post-baseline), as well as partner outcomes. The investigators will evaluate possible mechanisms of change including partner support and individual and partner motivation to quit as well as evaluate the cost and relative cost of each abstainer within and across condition. These data on the efficacy, mechanisms, and costs of FITs for DSCs will inform population level implementation and promote successful quitting in this treatment refractory population.

DETAILED DESCRIPTION:
The proposed study investigates the efficacy of implementing Financial Incentivized Treatments (FITs) in dyads on smoking abstinence in DSCs. The core design is a three-group longitudinal design in which participants are randomized into one of three conditions (no-FIT control, SFIT (one couple member offered incentives) and DFIT (both couple members offered incentives and tracked across 12 months. During this time, participants will complete a baseline session, be offered quitting resources (e.g. psychoeducation, NRT), and complete four follow-ups (1, 3, 6 [primary efficacy timepoint], and 12 months scheduled post-baseline). In all conditions, all participants (both targets and partners) will receive combination fast- and slow-acting NRT (calibrated to their smoking heaviness and/or time to first cigarette) and access to quitting resources.

In all conditions, the target will be determined as the first person to make contact with the research team in response to study advertising. The investigators estimate 70% of targets will be female. The investigators will stratify to create approximately equal proportions of target sex by cell. Same sex couples will be independently stratified across conditions to attempt to balance proportionate representation (estimated prevalence of same sex couples = 8%). Because heaviness of smoking (<20 vs 20+ cigarettes/day) requires a different NRT regimen and heaviness of smoking is associated with different quit rates, the investigators will also stratify random assignment based on number of cigarettes per day. Collectively, these strategies will enhance the likelihood of equivalent composition by condition.

Targets will be randomly assigned to one of three conditions. Consistent with the R21 design, participants in the no-FIT control condition will not receive incentives. Targets in the SFIT condition will be offered financial incentives for biochemically verified abstinence ($200 at each of three follow-ups [1, 3, and 6 Month]). In the DFIT condition, both targets and partners will be offered financial incentives for abstinence. Thus, in this condition, the total financial incentives offered to the dyad are twice the amount as offered to participants in the SFIT condition. However, because partners are involved in learning about the incentives, partner involvement is relatively high in both conditions. Partner involvement and understanding of the situation will be assessed as a potential mechanism of FIT efficacy. This design extends our pilot study to examine the efficacy of FITs for long-term abstinence and then then examines whether offering incentives to both members adds additional benefit beyond offering incentives to one member of the couple.

A total of 450 DSC targets (900 total smokers) will be recruited from across the United States. In all conditions, the target will be determined as the first person to contact the research team in response to study advertising. Couples will be defined as two people involved in a romantic relationship for at least 6 months who are married or cohabiting. Inclusion criteria are: 1) age of 18+; 2) smoking of 5+ cigarettes/day; 3) relationship status of married to or living with a daily smoker of 5+ cigarettes who is also above the age of 18; and 4) romantic Exclusion criteria are: 1) less than 8th grade capacity to read and write in English; 2) recent hospitalization (past 6 months) 3) psychosis risk; 4) regular (4+ days weekly) use of e-cigarettes; 5) Contra-indication for NRT (e.g., pregnancy, heart disease); 6) Marijuana use. Inclusion and exclusion criteria apply to both members of each couple; both members of each couple must be eligible for the target to enroll. Inclusion and exclusion criteria apply to both members of each couple. Study participation will last 1 year, including an initial Baseline session, three incentivized follow-ups (1 Mth, 3 Mth, 6 Mth follow-ups) and an unincentivized follow-up (12 Mth). Both members of each couple will be assessed at each time point, regardless of condition. Assessments will be completed by targets and partners via remote video conference at Baseline, 1 Mth, 3 Mth, 6 Mth, and 1 year. The investigators will measure smoking history, point-prevalence abstinence, heaviness of smoking, nicotine dependence, and possible motivational and dyadic mechanisms and moderators of anticipated effects.

ELIGIBILITY:
Inclusion Criteria:

* 1) age of 18+; 2) smoking of 5+ cigarettes/day; 3) relationship status of married to or living with a daily smoker of 5+ cigarettes who is also above the age of 18; and 4) romantic relationship duration of at least six months.

Exclusion Criteria:

* 1) less than 8th grade capacity to read and write in English; 2) recent hospitalization (past 6 months) 3) psychosis risk; 4) regular (4+ days weekly) use of e-cigarettes; 5) Contra-indication for NRT (e.g., pregnancy, heart disease); 6) Marijuana use.

Inclusion and exclusion criteria apply to both members of each couple; both members of each couple must be eligible for the target to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Point-Prevalence Abstinence at End of Treatment | 6 Month
  % of targets (intent to treat sample) who are abstinent (self-report no smoking past 7 days + expired carbon monoxide (CO) <= 5 ppm

SECONDARY OUTCOMES:
Point-Prevalence Abstinence After Treatment | 1 year
  % of targets (intent to treat sample) who are abstinent (self-report no smoking past 7 days + expired CO <= 5 ppm
Point-Prevalence Abstinence at First Follow-up | 1 month
  % of targets (intent to treat sample) who are abstinent (self-report no smoking past 7 days + expired CO <= 5 ppm
Point-Prevalence Abstinence at Second Follow-up | 3 month
  % of targets (intent to treat sample) who are abstinent (self-report no smoking past 7 days + expired CO <= 5 ppm
Partner Point-Prevalence Abstinence | 1 Month, 3 Month, 6 Month, 1 Year
  % of partners (intent to treat sample) who are abstinent (self-report no smoking past 7 days + expired CO <= 5 ppm at each follow-up
Smoking Heaviness | 1 Month, 3 Month, 6 Month, 1 Year
  All participants will report their average daily cigarette consumption at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R vanDellen, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared including key study variables (predictors and outcomes) through Open Science Framework (OSF).
Supporting Information: ICF
Time Frame: Individual participant data (IDP) will become available 6 months after publication or August 2029, whichever comes later.
Access Criteria: To protect participant anonymity, some identifying information will only be available through coordination with the study principal investigator (PI) (e.g., gender, same sex status, age, race).

REFERENCES:
- [Background] vanDellen MR, Wright JWC, Zhao B, Cullinan C, Beach SRH, Shen Y, Haskins LB, Schiavone WM, MacKillop JM. Partner-Involved Financial Incentives for Smoking Cessation in Dual-Smoker Couples: A Randomized Pilot Trial. Nicotine Tob Res. 2024 Jan 22;26(2):229-236. doi: 10.1093/ntr/ntad183. PMID 37742229

DOCUMENTS (1):
  • Informed Consent Form (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT06296849/ICF_000.pdf